CLINICAL TRIAL: NCT03184363
Title: Efficacy and Safety of DWP450 for Treating Crows Feet Lines(CFL) in Combination With Glabellar Lines: Multi-center, Single Arm, Open, Extension Study
Brief Title: Efficacy and Safety of DWP450 for Treating Crows Feet Lines(CFL) in Combination With Glabellar Lines(Extension Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP450005E
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Crow's Feet Lines; Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clostridium Botulinum A Toxin (Experimental): Clostridium Botulinum A Toxin
  Interventions: Drug: Clostridium Botulinum A Toxin

INTERVENTIONS:
Drug: Clostridium Botulinum A Toxin — Clostridium Botulinum A Toxin

SUMMARY:
The purpose of this study is to explore the Efficacy and Safety of DWP450 for treating Crows Feet Lines(CFL) in combination with glabellar line(GL) as extension study of phase 3 study for CFL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 18 to 75 years old
* moderate-to-severe CFL at maximum smile on the FWS as rated by the investigator
* moderate-to-severe GL at maximum frawn on the FWS as rated by the investigator
* Subject who has completed phase 3 study for CFL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Subject Assessment of Satisfaction of Appearance | At 4 weeks
  Subject Assessment of Satisfaction of Appearance

IPD SHARING:
Plan to Share IPD: Undecided